CLINICAL TRIAL: NCT05160857
Title: Clinical Study on the Efficacy and Safety of Hetropapa Ethanolamine Tablets in the Treatment of Thrombocytopenia Caused by Concurrent Radiotherapy and Chemotherapy in Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Wu jin rong, researcher, Second Hospital of Shanxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SecondShanxiMU
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Tumor Chemotherapy-related Thrombocytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test group (Experimental)
  Interventions: Drug: Herombopag Olamine

INTERVENTIONS:
Drug: Herombopag Olamine — The initial dose of hetropapa is recommended to be 7.5mg, once a day, oral on an empty stomach, and can only be eaten after oral administration for 2 hours, so as to avoid taking it with meals.

SUMMARY:
This study is a single arm, single center and exploratory clinical study, which aims to explore the efficacy and safety of hetropapa ethanolamine tablets in the treatment of thrombocytopenia caused by concurrent radiotherapy and chemotherapy of cervical cancer. The primary end point was the proportion of subjects who were effective after treatment with hetropapa in the first cycle after treatment, that is, the platelet value recovered to ≥ 100 x 109 / L after treatment. The main inclusion criteria were: voluntary participation in the trial and signing informed consent; Age ≥ 18 years old, regardless of gender; Cervical cancer was diagnosed by histopathology or cytology; Platelet < 75 × 109/L； At the time of screening, the expected survival time is ≥ 12 weeks, and can be treated with the current chemotherapy regimen for at least 1 cycle.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the trial and sign the informed consent form; Age ≥ 18 years old, regardless of gender; Cervical cancer was diagnosed by histopathology or cytology; Platelet < 75 × 109/L At the time of screening, the expected survival time is ≥ 12 weeks, and can be treated with the current chemotherapy regimen for at least 1 cycle

Exclusion Criteria:

* Screening or baseline platelet value < 30 × 109/L Suffering from the following hematopoietic system diseases other than thrombocytopenia (CIT) caused by tumor chemotherapy drugs, including but not limited to leukemia, primary immune thrombocytopenia, bone marrow proliferative diseases, multiple myeloma and myelodysplastic syndrome; Thrombocytopenia caused by causes other than CIT occurred within 6 months before screening, including but not limited to chronic liver disease, hypersplenism, infection and bleeding; Clinical manifestations of severe bleeding within 2 weeks before screening, such as gastrointestinal tract or central nervous system bleeding; Neutrophil absolute value < 1.0 × 109 / L, hemoglobin < 80g / L; It is allowed to use granulocyte colony stimulating factor, erythrocyte and EPO infusion in line with clinical routine; The researcher believes that participating in the trial has a great risk to the subject's health or safety, or other situations that may affect the efficacy evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet index | Blood routine tests were conducted every three days within 14 days after taking the drug
  Destroy after use

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No